CLINICAL TRIAL: NCT05916378
Title: Achieving Equity in Genomic Testing for Breast Cancer Through Partner-Led Strategies and Policies
Status: Active, not recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: The Latino Cancer Institute (Unknown)
Responsible Party: Principal Investigator, Manali Indravadan Patel, Principal Investigator, Stanford University
Other Study IDs: 68742
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: Genomic Testing; Precision Breast Cancer Care; Precision Medicine
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients and Caregivers: We will survey 100 patients and 50 caregivers.

SUMMARY:
The purpose of this study is to identify the barriers, and the extent of said barriers, to genomic testing for breast cancer patients among low-income and minority populations, particularly throughout Northern California. The investigators have created a survey that is available online for any patient with cancer to fill out voluntarily regarding their experiences to date. The survey is available at: https://stanforduniversity.qualtrics.com/jfe/form/SV_7VElf8oesWcB3bE

DETAILED DESCRIPTION:
The study has two main data-collecting phases. In phase 1, the investigators will engage multilevel stakeholders to respond to a survey assessing experience with and perceptions of genomic testing and its accessibility for patients with breast cancer in California. In phase 2, selected and interested survey participants who voluntarily provide their contact information on the survey will be asked to participate in an in-depth 1:1 semi-structured interview to explore disparities in genomic testing for breast cancer more closely. The investigators will then utilize their findings from both phases to present aggregate findings to an Expert Panel and Community Advisory Board and work together to develop policy recommendations. The policy recommendations will then be presented to policy makers, with the aim of identifying sustainable solutions that address breast cancer treatment and outcome disparities throughout Northern California.

ELIGIBILITY:
Inclusion Criteria:

* The patients must be 18 years or older.
* Patients who opt in to complete the survey.
* Patients must have the capacity to verbally consent for the interview.

Exclusion Criteria:

* Patients who under the age of 18 years old.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We expect to recruit 150 participants for enrollment in phase 1. These participants will include 100 patients diagnosed with breast cancer and 50 caregivers. In phase 2, we expect to recruit 55 of our phase 1 survey participants to complete a one-time one-on-one in-depth interview.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who fill out the survey and participate in the semi-structured interviews. [ Time Frame: 12 Months ] | 12 Months
  We will track the number of participants who fill out the survey for the 12 month duration of the study and the number of participants who participate in the semi-structured telephone interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT05916378/ICF_001.pdf